CLINICAL TRIAL: NCT05593081
Title: Multicenter Study of Fulminant Type 1 Diabetes in China
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, professor, Second Xiangya Hospital of Central South University
Other Study IDs: F1 China
Record Dates: First submitted 2022-10-18; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes: HLA ; fulminant
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: HLA — Distinguish based on clinical features

SUMMARY:
This study took FT1D（fulminant type 1 diabetes） as the research object, collected the cases of FT1D patients, and described the clinical characteristics of this type of disease. The HLA susceptibility genes of FT1D were identified by PCR and other techniques, taking age-sex-matched healthy subjects as controls and HLA genes as the research entry point.

DETAILED DESCRIPTION:
1. FT1D cases related to different etiologies were collected. The collected case data were the clinical data at the time of hospitalization for the first episode of FT1D, including the history of present illness, past history, vital signs, blood glucose at the onset, blood gas analysis, myocardial enzymes, pancreatic enzymes, glycosylated hemoglobin, C Peptides, islet autoantibodies and other laboratory indicators. Analysis and research are carried out according to factors such as the pathogenesis of the patients, so as to conduct a complete analysis of the pathogenesis characteristics of such patients under the condition of expanding cases, so as to improve the understanding of the disease and the level of diagnosis and treatment of the disease.
2. The study collected 240 patients in the FT1D group and 250 patients in the control group with genetic blood (previous research has been available), analyzed the HLA gene, and compared the risk and frequency of HLA class II alleles, genotypes and haplotypes between the two groups. , to explore the susceptibility risk genes and protective properties of Chinese FT1D patients. According to GADA positive and negative, the comparison of the susceptibility of Chinese FT1D class II HLA genotype, from the perspective of genetics to explore the role of antibodies in the pathogenesis of FT1D.

ELIGIBILITY:
patients with fulminant 1 diabetes

Inclusion Criteria:

1) diabetic ketosis or ketoacidosis occurred soon after the onset of hyperglycemic symptoms; 2) patient presented with plasma glucose ≥16.0 mmol/L and HbA1c <8.7% at the first visit; and 3) patient had urinary C-peptide excretion <10 µg/day,fasting serum C-peptide level <0.10 nmol/L, or postprandial serum C-peptide <0.17 nmol/L at onset

Exclusion Criteria:

Case reports of previously diagnosed with diabetes were excluded.

Healthy Volunteers

Inclusion Criteria:

* Normal control: The inclusion criteria are as follows: (1) Oral glucose tolerance test (OGTT): fasting blood glucose (FPG) <5.6 mmol/L and postprandial 2 h blood glucose (PPG) <7.8 mmol/L. The participants voluntarily signed the informed consent and extracted 3ml of peripheral blood for DNA extraction.

Exclusion Criteria:

* The exclusion criteria were as follows: (1) with heart, brain, liver, kidney or other chronic diseases; (2) with other types of autoimmune diseases; (3) with malignant tumors; (4) with a family history of diabetes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with fulminant 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum hemoglobin A1c level | Every year for up to 5 years
  A1c reflects the average blood glucose level

SECONDARY OUTCOMES:
Change in titer of autoantibodies | Every year for up to 5 years
  Glutamic acid decarboxylase antibody
Treatment options | Every year for up to 5 years
  Insulin use protocol and total amount
The incidence of chronic complications of diabetes mellitus | up to 5 years
  The incidence of diabetic neuropathy, diabetic nephropathy and diabetic retinopathy

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Quanzhou First People's Hospital, Quanzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Zunyi, Guangzhou
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Changsha Central Hospital, Changsha, Hunan
  - Yancheng Third People's Hospital, Yancheng, Jiangs
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Yunnan Provincial People's Hospital, Kunming, Yunnan
  - The Second Xiangya Hospital of Central South University, Changsha

IPD SHARING:
Plan to Share IPD: No